CLINICAL TRIAL: NCT00876174
Title: Effects of Genotypes on Interferon Signaling in Chronic Hepatitis C
Status: Withdrawn | Type: Observational
Why Stopped: no accrual
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0143-09-EP
Record Dates: First submitted 2009-04-02; First posted 2009-04-06 (Estimated); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; Genotype 1
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 20 ml blood for peripheral mononuclear cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: 20 patients with genotype 1, chronic hepatitis C who are to undergo standard antiviral therapy
  Interventions: Procedure: Blood sampling of peripheral blood mononuclear cells
- control: Group 2, (control): 10 healthy family members or significant others of patients who are to undergo standard antiviral therapy
  Interventions: Procedure: Blood draw, 20ml peripheral blood mononuclear cells

INTERVENTIONS:
Procedure: Blood sampling of peripheral blood mononuclear cells — Group 1, (Patients): PMBC (20 ml blood) to be drawn at baseline, weeks 4 and 12 during antiviral therapy and 24 weeks following the end of antiviral therapy
  Groups: Patients
Procedure: Blood draw, 20ml peripheral blood mononuclear cells — One time blood draw of 20 ml
  Groups: control

SUMMARY:
The objective of this pilot project is to investigate the prognostic criteria for sensitivity of Chronic Hepatitis C (CHC) Genotype 1, patients to IFNa treatment. Signal transduction in peripheral blood mononuclear cell (PBMC) of control groups will be compared with that of CHC patients. For this study, 20 patients with Hepatitis C virus (HCV) infection who are to undergo standard antiviral therapy and 10 healthy donors (significant others of the HCV subject) will be enrolled. Signal transduction will be studied in peripheral blood of CHC subjects before the treatment, after 1 and 3 months of treatment, and 4-6 months following the completion of treatment.

DETAILED DESCRIPTION:
In addition, the mechanism of non-responsiveness of HCV patients to IFNa will be studied. For this purpose, formation of complexes between STAT1 and its negative regulator, PIAS1 (immunoprecipitation, Western blot) will be examined. In comparing subjects on standard therapy vs the addition of betaine, (under separate studies) we will assess whether the formation of STAT1-PIAS1 complexes is due to impaired methylation on STAT1 on arginine residues which may be over come by the addition of betaine.

ELIGIBILITY:
Inclusion Criteria

* 19 years of age or older, of either gender
* History of chronic hepatitis C documented by HCVRNA or healthy family member/significant other
* Documented genotype 1 for hepatitis participants or no hepatitis infection for healthy control
* Subject prescribed antiviral therapy for hepatitis participants or none for healthy control
* Able to give informed consent

Exclusion Criteria

* Under 19 years of age
* Unable to give informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with genotype 1, chronic hepatitis C who are to undergo antiviral therapy and their healthy family member or significant other
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-04-15 (Actual); Primary Completion 2010-01-08 (Actual); Study Completion 2010-01-08 (Actual)

PRIMARY OUTCOMES:
Prognostic criteria for sensitivity of Chronic Hepatitis C patients to interferon alpha treatment | 3 years
  To investigate the prognostic criteria for sensitivity of Chronic Hepatitis C patients to interferon alpha treatment

SECONDARY OUTCOMES:
Effects of antiviral treatment on interferon gene signaling in peripheral blood mononuclear cells | 3 years
  To determine the effects of antiviral treatment on interferon gene signaling in peripheral blood mononuclear cells

CONTACTS AND LOCATIONS:
Overall Officials: Mark E Mailliard, MD, Principal Investigator — University of Nebraska